CLINICAL TRIAL: NCT00886769
Title: A Randomized, Double-blind, Placebo Controlled, Single-dose Study to Assess the Initial Efficacy of Canakinumab (ACZ885) With Respect to the Adapted ACR Pediatric 30 Criteria in Patients With Systemic Juvenile Idiopathic Arthritis (SJIA) and Active Systemic Manifestations
Brief Title: Single-dose Study to Assess Efficacy of Canakinumab (ACZ885) in Patients With Active Juvenile Idiopathic Arthritis (SJIA)
Acronym: β-SPECIFIC 1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recommendation by Data Monitoring Committee
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network); Southwest Pediatric Nephrology Study Group (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885G2305; EudraCT: 2008-005476-27
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Systemic Juvenile Idiopathic Arthritis
Keywords: Flare; arthritis; IL-1beta antagonist; systemic juvenile idiopathic arthritis; Juvenile Rheumatoid; Systemic juvenile idiopathic arthritis with active flare
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Canakinumab (Experimental): Patients received a single dose of subcutaneous(sc) injection of canakinumab (4 mg/kg) on Day 1. Maximal total single dose of canakinumab allowed was 300 mg. Any patient who required a dose greater than 150 mg (patients>37.5 kg) received two sc injections.
  Interventions: Drug: Canakinumab
- Placebo (Placebo Comparator): Patients received a single dose matching placebo of canakinumab on day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab — Canakinumab was supplied in individual 6 mL glass vials each containing 150 mg canakinumab powder as a lyophilized cake. Each reconstituted vial provided 150mg of canakinumab per 1 mL.
  Other Names: ACZ885
  Arms: Canakinumab
Drug: Placebo — Placebo was provided in individual 6 mL glass vials each containing 150 mg placebo powder matching canakinumab as a lyophilized cake. Each reconstitued vial provided 150mg of placebo per 1 mL.
  Arms: Placebo

SUMMARY:
This study assessed the initial efficacy and safety of canakinumab over a 4 week period in patients with systemic juvenile idiopathic arthritis (SJIA) having a flare. Response to treatment will be according to the adapted American College of Rheumatology(ACR)Pediatric 30 criteria at Day 15.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of systemic juvenile idiopathic arthritis as per ILAR definition that must have occurred at least 2 months prior to enrollment with onset of disease < 16 years of age:

   * Arthritis in one or more joints with or preceded by fever of at least 2 weeks duration that is documented to be daily/quotidian for at least 3 days and accompanied by one or more of the following:
   * evanescent nonfixed erythematous rash,
   * generalized lymph node enlargement,
   * hepatomegaly and/ or splenomegaly,
   * serositis
2. Parent's or legal guardian's written informed consent and child's assent, if appropriate, or patient's informed consent for ≥ 18 years of age
3. Male and female patients aged ≥ 2 to < 20 years of age
4. Active disease at the time of enrollment defined as follows:

   * At least 2 joints with active arthritis
   * Documented spiking, intermittent fever (body temperature > 38°C) for at least 1 day during the screening period within 1 week before first canakinumab/placebo dose
   * C-reactive protein (CRP) > 30 mg/L (normal range < 10 mg/L)
5. Naïve to canakinumab
6. Other protocol defined inclusion criteria may apply

Exclusion Criteria:

Patients who fulfilled one or more of the following criteria were not eligible for inclusion in this study:

1. Pregnant or nursing (lactating) female patients
2. Female patients having reached sexual maturity unless their career, lifestyle, or sexual orientation precluded intercourse with a male partner and/or they were using an acceptable method of contraception
3. History of hypersensitivity to study drug or to biologics.
4. Diagnosis of active macrophage-activation syndrome (MAS) (Ravelli, Magni-Manzoni and Pistorio 2005) within the last 6 months
5. With active or recurrent bacterial, fungal or viral infection, including patients with evidence of human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C infection
6. Other protocol defined exclusion criteria may apply

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (91):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital Research Inst, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Tufts New England Medical Center-Dept. of Allergy, Boston, Massachusetts
  - St. Barnabas Ambulatory Care Center, Livingston, New Jersey
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital/Neurology, Cinncinati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Legacy Emanuel Hospital, Portland, Oregon
  - Legacy Emanual Research, Portland, Oregon
  - Specially For Children, Austin, Texas
- Argentina (3):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Capital Federal
  - Novartis Investigative Site, La Plata
- Belgium (4):
  - Novartis Investigative site, Brussels
  - Novartis Investigative site, Ghent
  - Novartis Investigative Site, Laken
  - Novartis Investigative site, Leuven
- Brazil (4):
  - Novartis Investigative Site, Curitiba
  - Novartis Investigative site, Porto Alegre
  - Novartis Investigative site, Rio de Janeiro
  - Novartis Investigative site, São Paulo
- Canada (5):
  - Novartis Investigative site, Vancouver, British Columbia
  - Novartis Investigative site, Halifax, Nova Scotia
  - Novartis Investigative site, Toronto, Ontario
  - Novartis Investigative site, Montreal, Quebec
  - Novartis Investigative site, Calgary
- Novartis Investigative site, Arhus N, Denmark
- France (4):
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
- Germany (15):
  - Novartis Investigative Site, Bad Bamstedt
  - Novartis Investigative site, Berlin
  - Novartis Investigative Site, Bremen
  - Novartis Investigative site, Dresden
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative site, Garmisch-Partenkirch
  - Novartis Investigative Site, Geißen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative site, Hanover
  - Novartis Investigative site, Krefeld
  - Novartis Investigative site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Saint Augustin
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative site, Tübingen
- Novartis Investigative site, Thessaloniki, Greece
- Novartis Investigative Site, Budapest, Hungary
- Israel (5):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
- Italy (9):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Genova
  - Novartis Investigative site, Milan
  - Novartis Investigative site, Napoli
  - Novartis Investigative site, Padua
  - Novartis Investigative site, Rome
  - Novartis Investigative site, Scafati
  - Novartis Investigative site, Torino
- Novartis Investigative site, Utrecht, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Lima, Peru
- Novartis Investigative site, Warsaw, Poland
- South Africa (3):
  - Novartis Investigative site, Berea, Durban
  - Novartis Investigative site, Mayville, Durban
  - Novartis Investigative site, Pretoria
- Spain (3):
  - Novartis Investigative site, Barcelona
  - Novartis Investigative site, Madrid
  - Novartis Investigative site, Valencia
- Novartis Investigative site, Stockholm, Sweden
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative site, Lausanne
  - Novartis Investigative site, Zurich
- Turkey (Türkiye) (3):
  - Novartis Investigative site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (7):
  - Novartis Investigative site, Birmingham
  - Novartis Investigative site, Liverpool
  - Novartis Investigative site, London
  - Novartis Investigative site, Manchester
  - Novartis Investigative site, New Castle Upon Tyne
  - Novartis Investigative site, Norwich
  - Novartis Investigative site, Oxford

REFERENCES:
- [Derived] Ruperto N, Brunner HI, Quartier P, Constantin T, Wulffraat NM, Horneff G, Kasapcopur O, Schneider R, Anton J, Barash J, Berner R, Corona F, Cuttica R, Fouillet-Desjonqueres M, Fischbach M, Foster HE, Foell D, Radominski SC, Ramanan AV, Trauzeddel R, Unsal E, Levy J, Vritzali E, Martini A, Lovell DJ; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Canakinumab in patients with systemic juvenile idiopathic arthritis and active systemic features: results from the 5-year long-term extension of the phase III pivotal trials. Ann Rheum Dis. 2018 Dec;77(12):1710-1719. doi: 10.1136/annrheumdis-2018-213150. Epub 2018 Sep 29. PMID 30269054
- [Derived] Brachat AH, Grom AA, Wulffraat N, Brunner HI, Quartier P, Brik R, McCann L, Ozdogan H, Rutkowska-Sak L, Schneider R, Gerloni V, Harel L, Terreri M, Houghton K, Joos R, Kingsbury D, Lopez-Benitez JM, Bek S, Schumacher M, Valentin MA, Gram H, Abrams K, Martini A, Lovell DJ, Nirmala NR, Ruperto N; Pediatric Rheumatology International Trials Organization (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Early changes in gene expression and inflammatory proteins in systemic juvenile idiopathic arthritis patients on canakinumab therapy. Arthritis Res Ther. 2017 Jan 23;19(1):13. doi: 10.1186/s13075-016-1212-x. PMID 28115015
- [Derived] Grom AA, Ilowite NT, Pascual V, Brunner HI, Martini A, Lovell D, Ruperto N; Paediatric Rheumatology International Trials Organisation and the Pediatric Rheumatology Collaborative Study Group; Leon K, Lheritier K, Abrams K. Rate and Clinical Presentation of Macrophage Activation Syndrome in Patients With Systemic Juvenile Idiopathic Arthritis Treated With Canakinumab. Arthritis Rheumatol. 2016 Jan;68(1):218-28. doi: 10.1002/art.39407. PMID 26314396
- [Derived] Ruperto N, Brunner HI, Quartier P, Constantin T, Wulffraat N, Horneff G, Brik R, McCann L, Kasapcopur O, Rutkowska-Sak L, Schneider R, Berkun Y, Calvo I, Erguven M, Goffin L, Hofer M, Kallinich T, Oliveira SK, Uziel Y, Viola S, Nistala K, Wouters C, Cimaz R, Ferrandiz MA, Flato B, Gamir ML, Kone-Paut I, Grom A, Magnusson B, Ozen S, Sztajnbok F, Lheritier K, Abrams K, Kim D, Martini A, Lovell DJ; PRINTO; PRCSG. Two randomized trials of canakinumab in systemic juvenile idiopathic arthritis. N Engl J Med. 2012 Dec 20;367(25):2396-406. doi: 10.1056/NEJMoa1205099. PMID 23252526
- See also: Click here for more information about this study — http://www.NovartisClinicalTrials.com
- See also: Related Info — http://www.juvenilearthritisresearch.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Canakinumab | Placebo
Started | 43 | 41
Completed | 37 | 4
Not Completed | 6 | 37
Not completed — Unsatisfactory therapeutic effect | 6 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab | Placebo | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (5.08) | 9.7 (4.32) | 9.0 (4.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Meet the Adapted American College of Rheumatology (ACR) Pediatric 30 Criteria
Description: Adapted ACR Pediatric 30 criteria determined responders (improved from baseline of at least 30% in at least 3 response variables 1-6 and no intermittent fever in preceding week [variable 7], with no more than one variable 1-6 worsening > 30% ) 1. Physician's Global Assessment of disease activity: 0-100 mm VAS 2.Parent/Patient's Global Assessment of Patient's overall wellbeing: 0-100mmVAS in Child Health Assessment Questionnaire (CHAQ) 3. Functional ability: CHAQ 4.Number of joints with active arthritis 5. Number of joints with limited of motion 6. Laboratory measure of inflammation CRP (mg/L)
Time Frame: Baseline, Day 15, Day 29
Population: The Full Analysis Set (FAS) consisted of all randomized patients who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 43 | 41
percentage of participants
  Day 15 | 83.7 | 9.8
  Day 29 | 79.1 | 9.8

2. Secondary Outcome: Percentage of Patients Achieving the Adapted ACR Pediatric 50 Criteria
Description: Adapted ACR Pediatric 50 criteria determined responders (improved from baseline of at least 50% in at least 3 response variables 1-6 and no intermittent fever in preceding week [variable 7], with no more than one variable 1-6 worsening > 30%) 1. Physician's Global Assessment of disease activity: 0-100 mm VAS 2. Parent/Patient's Global Assessment of Patient's overall wellbeing: 0-100mmVAS in Child Health Assessment Questionnaire (CHAQ) 3. Functional ability: CHAQ 4. Number of joints with active arthritis 5. Number of joints with limited of motion 6. Laboratory measure of inflammation CRP (mg/L)
Time Frame: Baseline, Day 15, Day 29
Population: The Full Analysis Set (FAS) consisted of all randomized patients who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 43 | 41
percentage of participants
  Day 15 | 67.4 | 4.9
  Day 29 | 76.7 | 4.9

3. Secondary Outcome: Percentage of Patients Achieving the Adapted ACR Pediatric 70
Description: Adapted ACR Pediatric 70 criteria determined responders (improved from baseline of at least 70% in at least 3 response variables 1-6 and no intermittent fever in preceding week [variable 7], with no more than one variable 1-6 worsening > 30% ) 1. Physician's Global Assessment of disease activity: 0-100 mm VAS 2. Parent/Patient's Global Assessment of Patient's overall wellbeing: 0-100mmVAS in Child Health Assessment Questionnaire (CHAQ) 3. Functional ability: CHAQ 4. Number of joints with active arthritis 5. Number of joints with limited of motion 6. Laboratory measure of inflammation CRP(mg/L)
Time Frame: Baseline, Day 15, Day 29
Population: The Full Analysis Set (FAS) consisted of all randomized patients who received at least one dose of study drug.
Measure: Number; unit: percent of participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 43 | 41
percent of participants
  Day 15 | 60.5 | 2.4
  Day 29 | 65.1 | 2.4

4. Secondary Outcome: Percentage of Patients Achieving the Adapted ACR Pediatric 90
Description: Adapted ACR Pediatric 90 criteria determined responders (improved from baseline of at least 90% in at least 3 response variables 1-6 and no intermittent fever in preceding week [variable 7], with no more than one variable 1-6 worsening > 30% ) 1. Physician's Global Assessment of disease activity: 0-100 mm VAS 2. Parent/Patient's Global Assessment of Patient's overall wellbeing: 0-100mmVAS in Child Health Assessment Questionnaire (CHAQ) 3. Functional ability: CHAQ 4. Number of joints with active arthritis 5. Number of joints with limited of motion 6. Laboratory measure of inflammation CRP(mg/L)
Time Frame: Baseline, Day 15, Day 29
Population: The Full Analysis Set (FAS) consisted of all randomized patients who received at least one dose of study drug.
Measure: Number; unit: percent of participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 43 | 41
percent of participants
  Day 15 | 41.9 | 0
  Day 29 | 46.5 | 2.4

5. Secondary Outcome: Percentage of Patients Achieving the Adapted ACR Pediatric 100
Description: Adapted ACR Pediatric 100 criteria determined responders (ie improved from baseline of at least 100% in at least 3 response variables 1-6 and no intermittent fever in preceding week [variable 7], with no more than one variable 1-6 worsening > 30% ) 1. Physician's Global Assessment of disease activity: 0-100 mm VAS 2. Parent/Patient's Global Assessment of Patient's overall wellbeing: 0-100mmVAS in Child Health Assessment Questionnaire (CHAQ) 3. Functional ability: CHAQ 4. Number of joints with active arthritis 5. Number of joints with limited of motion 6. Laboratory measure of inflammation
Time Frame: baseline, Day 15, Day 29
Population: The Full Analysis Set (FAS) consisted of all randomized patients who received at least one dose of study drug.
Measure: Number; unit: percent of participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 43 | 41
percent of participants
  Day 15 | 32.6 | 0
  Day 29 | 32.6 | 2.4

6. Secondary Outcome: Change in Patient's Pain Intensity as Assessed on a 100-mm Visual Analog Scale (VAS)as Part of the Childhood Health Assessment Questionnaire(CHAQ)
Description: CHAQ assessed physical ability and functional status of patients as well as quality of life. The disability dimension consisted of 20 multiple choice items about difficulty in doing eight common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and activities. Four response categories range from 'without any difficulty' (0) to 'unable to do' (3). The parent's or patient's pain assessment was on VAS that was part of CHAQ. The VAS scale ranges from no pain (0 mm) to very severe pain (100 mm). Negative change indicates improvement.
Time Frame: Baseline, Day 15
Population: The Full Analysis Set (FAS) consisted of all randomized patients who received at least one dose of study drug. Only observed cases were used in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 43 | 25
Units on a scale | 20.3 (5.08) | 66.7 (6.35)

7. Secondary Outcome: Change in Patient's Pain Intensity as Assessed on a 100-mm Visual Analog Scale (VAS) as Part of CHAQ
Description: CHAQ, assessed physical ability and functional status of patients as well as quality of life. The disability dimension consisted of 20 multiple choice items about difficulty in doing eight common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and activities. Four response categories range from 'without any difficulty'(0) to 'unable to do' (3). The parent's or patient's pain assessment was on VAS that was part of CHAQ. The VAS scale ranges from no pain (0 mm) to very severe pain (100 mm). Negative change indicates improvement.
Time Frame: Baseline, Day 29
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 38 | 7
Units on a scale | 20.6 (5.59) | 62.5 (9.7)

8. Secondary Outcome: Percentage of Patients Who Had Body Temperature ≤ 38°C
Description: Body temperature was derived from vital signs evaluation. No conversion of body temperature was performed, no matter how it was measured.
Time Frame: Day 3
Population: as for outcome 6
Measure: Number; unit: Percent of participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 43 | 38
Percent of participants | 100 | 86.8

9. Secondary Outcome: Change in Health-related Quality of Life (HRQoL)Over Time by Use of the Child Health Questionnaire - Parent Form (CHQ-PF50)
Description: CHQ-PF50 measures HRQoL in children 5-18 years old from parent's perspective. Questionnaire completed by parent without input from patient. Total score ranges from 0-100. Increases in scores represent improved well-being in subjects as assessed by their parents. Mixed linear model on change from baseline in CHQ-PF50 score with treatment group, stratification factors, day of assessment and interaction between group and day as covariates. Covariance analysis used a repeated measures approach, so all timepoints over time were taken into account.
Time Frame: Over 4 week study period (Baseline, Day 15, Day 29)
Population: The Full Analysis Set (FAS) consisted of all randomized patients who received at least one dose of study drug. Observed cases only were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 28 | 34
units on a scale
  CHQ-PF50 physical score | 16.9 (3.46) | 4.9 (3.97)
  CHQ-PF50 psychosocial score | 6.2 (2.15) | -1.1 (2.49)

10. Secondary Outcome: Change in Disability Score Over Time by Use of the CHAQ
Description: The disability dimension of CHAQ consisted of 20 multiple choice items about difficulty in doing eight common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and activities. Four response categories range from 'without any difficulty'(0) to 'unable to do' (3). Mixed linear model on change from baseline in CHAQ score included treatment group, stratification factors, day of assessment and interaction between group and day as covariates. Negative change indicates improvement.
Time Frame: At 4 week study period
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 43 | 41
Units on a Scale | -0.8 (0.15) | -0.2 (0.20)

ADVERSE EVENTS:
Arm/Group | Canakinumab | Placebo
Serious Adverse Events (participants affected / at risk) | 2/43 | 2/41
Other Adverse Events (participants affected / at risk) | 17/43 | 3/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=43) | Placebo (N=41)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=43) | Placebo (N=41)
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 2 | 0
Headache (Nervous system disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until publication of the pooled data (i.e., data from all sites) in the clinical trial or publication of trial results in their entirety.